CLINICAL TRIAL: NCT01283438
Title: A Prospective, Randomized, Multicenter Study to Demonstrate the Superiority of the Barricaid® to Discectomy for Primary Lumbar Disc Herniation: Extended Follow-Up of the Barricaid® Annular Closure Device (ACD) Randomized Control Trial (RCT) Postmarket Cohort for Lumbar Disc Herniation and Interaction With Other Risk Factors
Brief Title: A Prospective, Randomized, Multicenter Study to Demonstrate the Superiority of the Barricaid to Discectomy for Primary Lumbar Disc Herniation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUBARD-CP-011
Record Dates: First submitted 2011-01-06; First posted 2011-01-26 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Barricaid Device (Experimental): Intervention: Barricaid Device
  Interventions: Device: Barricaid
- Standard of Care (Active Comparator): Standard (Limited) Discectomy Only
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Barricaid — Annular closure device
  Arms: Barricaid Device
Device: Standard of Care — Standard Limited discectomy
  Arms: Standard of Care

SUMMARY:
A randomized study to demonstrate the superiority of the Barricaid® when used in conjunction with limited discectomy, compared to limited discectomy alone, with regard to preventing reherniation and the recurrence of pain or dysfunction.

DETAILED DESCRIPTION:
The Barricaid is indicated for patients with radiculopathy (with or without back pain), a positive Straight Leg Raise (L45, L5S1) or femoral stretch test (L12, L23, L34), and a posterior or posterolateral herniation at one level between L1 and S1 with radiographic confirmation of neural compression using MRI who are found to have an annular defect (post discectomy) which measures between 4mm and 6mm tall and between 6mm and 10mm wide, have a minimum posterior disc height of 5mm, and have failed at least 6 weeks of conservative treatment including a post-approval amendment with follow-up visits at 7 & 10 years for eligible subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years old and skeletally mature (male or female).
* Patients with posterior or posterolateral disc herniations at one level between L1 and S1 with radiographic confirmation of neural compression using Magnetic Resonance Imaging (MRI).
* At least six (6) weeks of failed, conservative treatment prior to surgery
* Oswestry Disability Index (ODI) Questionnaire score of at least 40/100 at baseline.
* Visual Analog Scale (VAS) leg pain (one or both legs) of at least 40/100 at baseline.
* Psychosocially, mentally and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

* Spondylolisthesis Grade II or higher (25% slip or greater).
* Prior surgery at the index lumbar vertebral level.
* Subject has scoliosis of greater than ten (10) degrees (both angular and rotational).
* Any metabolic bone disease.
* Subject has insulin-dependent diabetes mellitus.
* Subject has been diagnosed with active hepatitis, acquired immunodeficiency syndrome (AIDS), or Human immunodeficiency virus (HIV).
* Subject has been diagnosed with rheumatoid arthritis or other autoimmune disease.
* Subject has a known allergy to titanium, polyethylene or polyester materials.
* Any subject that cannot have a baseline MRI taken.
* Subject is pregnant or interested in becoming pregnant in the next three (3) years.
* Subject has active tuberculosis or has had tuberculosis in the past three (3) years.
* Subject is currently involved in another investigational study.
* Any contraindication for MRI or Computed tomography CT scan (e.g. claustrophobia, contrast allergy).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2010-12-17 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Combined success of multiple clinical outcomes, including Oswestry disability index, Visual Analog Scale (VAS), and multiple radiographically confirmed measures | 24 months
  To be considered a success, a patient will have achieved success in each of the following outcomes:
  * 15 point (out of 100 point scale) improvement in Oswestry compared to pre-op
  * 20 point (on a 100 point scale) improvement in VAS Leg (based on the primary leg complaint; if both legs have a minimum of 40/100 pre-operatively, the average leg score will be used)
  * Maintenance of average disc height (75% or greater of preoperative disc height) compared to pre-op
  * No deterioration of neurological status at the index level measured by motor function
  * Device integrity and lack of implant migration (radiographic, implanted patients only)
  * No radiographically confirmed spontaneous fusion
  * No radiographically or surgically confirmed reherniation at the index level (on either side)
  * No secondary surgical interventions at the index level
No radiographic evidence of recurrent disc herniation | 24 months
  To be considered a success, a patient will have no evidence of recurrent disc herniation at the index level at any time up to and including the 24-month follow-up. Recurrent herniation may be confirmed surgically, or radiographically as determined by an independent review (unless surgically confirmed that the suspected herniation is not a herniation, e.g. scar tissue or residual nucleus material).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Back Pain Improvement | 24 months
  Change in back pain as measured using a Visual Analog Scale (VAS), on a scale of 0-100, with lower values representing better outcome. A subject is a success if there is at least a 20 point improvement on the VAS back at 24 months, relative to baseline.
Oswestry Disability Index (ODI) Improvement | 24 months
  Change in function as measured using the Oswestry Disability Index (ODI). The ODI is scored on a scale from 0% to 100%, with higher scores indicating higher levels of disability. A subject is a success if there is at least a 15 point improvement (decrease) in the ODI at the 24 month visit relative to baseline.
Reoperation | 24 months
  A subject will be deemed a success if they have not had a second operation at the index level by the 24 month visit. Rates of subject success in treatment and control will be compared at 24 months. A subject is a success if there is at least 75% of the pre-op disc height preserved at the 24 month visit.
Visual Analog Scale (VAS) LEG Pain Improvement | 24 months
  Change in leg pain as measured using a Visual Analog Scale (VAS), on a scale of 0-100, with lower values representing better outcome. A subject is a success if there is at least a 20 point improvement on VAS leg pain in the ipsilateral leg at 24 months, relative to baseline.
Disc Height Maintenance | 24 months
  A subject is a success if there is at least 75% of the pre-op disc height preserved as measured on MRI, at the 24 month visit.

OTHER OUTCOMES:
Post 5Y device or procedure-related Serious Adverse Event (SAE) | Post 60 months
  Adverse events will be categorized as device-related and/or procedure-related and will be assigned severity or seriousness. Safety will be determined by evaluating the type, frequency, severity, and relationship to device and/or procedure of adverse events through the 10 year time point or until stabilization of the endplate lesions, whichever is longer.
Post 5Y secondary surgical intervention at the index level | Post 60 months
  The safety will be supported if the incidence of secondary surgical interventions (SSIs) and the incidence SAEs related to either the device or procedure is not greater in the Barricaid® annular closure device than in the Control cohort.

CONTACTS AND LOCATIONS:
Locations (21):
- Austria (2):
  - LKH Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
- Belgium (3):
  - OLV Aalst, Aalst
  - ZNA Middleheim / AZ Klina, Antwerp
  - AZ Nikolaas, Sint-Niklaas
- CHRU Lille, Hôpital Roger Salengro, Lille, France
- Germany (10):
  - Orthopädische Klinik und Poliklinik - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Neurochirurgische Universitätsklinik Knappschafts-Krankenhaus Bochum-Langendreer, Bochum, North Rhine-Westphalia
  - Klinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Deggendorf, Deggendorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Asklepios Westklinikum Hamburg, Hamburg
  - UNI Kiel, Kiel
  - St. Bonifatius Hospital GmbH, Lingen
  - UMM Mannheim, Mannheim
- Netherlands (4):
  - SLAZ Amsterdam, Amsterdam
  - MCH Antoniushove, Leidschendam
  - MCH Westeinde, The Hague
  - Isala Klinieken, Zwolle
- KSA Aarau, Aarau, Switzerland

REFERENCES:
- [Result] Thome C, Klassen PD, Bouma GJ, Kursumovic A, Fandino J, Barth M, Arts M, van den Brink W, Bostelmann R, Hegewald A, Heidecke V, Vajkoczy P, Frohlich S, Wolfs J, Assaker R, Van de Kelft E, Kohler HP, Jadik S, Eustacchio S, Hes R, Martens F; Annular Closure RCT Study Group. Annular closure in lumbar microdiscectomy for prevention of reherniation: a randomized clinical trial. Spine J. 2018 Dec;18(12):2278-2287. doi: 10.1016/j.spinee.2018.05.003. Epub 2018 May 3. PMID 29730458
- [Result] Martens F, Vajkoczy P, Jadik S, Hegewald A, Stieber J, Hes R. Patients at the Highest Risk for Reherniation Following Lumbar Discectomy in a Multicenter Randomized Controlled Trial. JB JS Open Access. 2018 Apr 16;3(2):e0037. doi: 10.2106/JBJS.OA.17.00037. eCollection 2018 Jun 28. PMID 30280130
- [Result] Klassen PD, Hsu WK, Martens F, Inzana JA, van den Brink WA, Groff MW, Thome C. Post-lumbar discectomy reoperations that are associated with poor clinical and socioeconomic outcomes can be reduced through use of a novel annular closure device: results from a 2-year randomized controlled trial. Clinicoecon Outcomes Res. 2018 Jun 26;10:349-357. doi: 10.2147/CEOR.S164129. eCollection 2018. PMID 29983583
- [Result] Ament J, Thaci B, Yang Z, Kulubya E, Hsu W, Bouma G, Kim KD. Cost-effectiveness of a Bone-anchored Annular Closure Device Versus Conventional Lumbar Discectomy in Treating Lumbar Disc Herniations. Spine (Phila Pa 1976). 2019 Jan 1;44(1):5-16. doi: 10.1097/BRS.0000000000002746. PMID 29927860
- [Result] Kursumovic A, Kienzler JC, Bouma GJ, Bostelmann R, Heggeness M, Thome C, Miller LE, Barth M; Annular Closure RCT study group. Morphology and Clinical Relevance of Vertebral Endplate Changes Following Limited Lumbar Discectomy With or Without Bone-anchored Annular Closure. Spine (Phila Pa 1976). 2018 Oct 15;43(20):1386-1394. doi: 10.1097/BRS.0000000000002632. PMID 29538243
- [Result] Klassen PD, Bernstein DT, Kohler HP, Arts MP, Weiner B, Miller LE, Thome C. Bone-anchored annular closure following lumbar discectomy reduces risk of complications and reoperations within 90 days of discharge. J Pain Res. 2017 Aug 26;10:2047-2055. doi: 10.2147/JPR.S144500. eCollection 2017. PMID 28894388
- [Derived] Thome C, Kursumovic A, Klassen PD, Bouma GJ, Bostelmann R, Martens F, Barth M, Arts M, Miller LE, Vajkoczy P, Hes R, Eustacchio S, Nanda D, Kohler HP, Brenke C, Fluh C, Van de Kelft E, Assaker R, Kienzler JC, Fandino J; Annular Closure RCT Study Group. Effectiveness of an Annular Closure Device to Prevent Recurrent Lumbar Disc Herniation: A Secondary Analysis With 5 Years of Follow-up. JAMA Netw Open. 2021 Dec 1;4(12):e2136809. doi: 10.1001/jamanetworkopen.2021.36809. PMID 34882183
- [Derived] Kienzler JC, Fandino J, Van de Kelft E, Eustacchio S, Bouma GJ; Barricaid(R) Annular Closure RCT Study Group. Risk factors for early reherniation after lumbar discectomy with or without annular closure: results of a multicenter randomized controlled study. Acta Neurochir (Wien). 2021 Jan;163(1):259-268. doi: 10.1007/s00701-020-04505-4. Epub 2020 Oct 21. PMID 33085021
- [Derived] van den Brink W, Fluh C, Miller LE, Klassen PD, Bostelmann R. Lumbar disc reherniation prevention with a bone-anchored annular closure device: 1-year results of a randomized trial. Medicine (Baltimore). 2019 Nov;98(44):e17760. doi: 10.1097/MD.0000000000017760. PMID 31689835
- [Derived] Kienzler JC, Klassen PD, Miller LE, Assaker R, Heidecke V, Frohlich S, Thome C; Annular Closure RCT Study Group. Three-year results from a randomized trial of lumbar discectomy with annulus fibrosus occlusion in patients at high risk for reherniation. Acta Neurochir (Wien). 2019 Jul;161(7):1389-1396. doi: 10.1007/s00701-019-03948-8. Epub 2019 May 15. PMID 31089894
- See also: Sponsor website — http://www.barricaid.com
- See also: Published protocol design manuscript — http://www.ijclinicaltrials.com/index.php/ijct/article/view/137/84